CLINICAL TRIAL: NCT06253377
Title: Exploring Clinical Management and Outcomes of Continuous Renal Replacement Therapy With Oxiris in Acute Kidney Injury and Sepsis
Brief Title: Continuous Renal Replacement Therapy With Oxiris in Acute Kidney Injury and Sepsis
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Nefro Consultoria de Doenças Renais Ltda (Network)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: Nefro01
Record Dates: First submitted 2023-12-10; First posted 2024-02-12 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2023-12

CONDITIONS: Acute Kidney Injury; Sepsis
Keywords: Acute Kidney Injury; Blood Purification; Adsorptive membranes; Sepsis; Cytokines
MeSH Terms: conditions — Acute Kidney Injury; Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Study cohort: Patients with Acute Kidney Injury and Renal Replacement Therapy indication, following local clinical patterns, who were treated with Continuous Renal Replacement Therapy with the adsorption membrane filter Oxiris™
  Interventions: Device: Adsorption membrane filter Oxiris™

INTERVENTIONS:
Device: Adsorption membrane filter Oxiris™ — Continuous Renal Replacement Therapy with the adsorption membrane filter Oxiris™

SUMMARY:
It is an epidemiology study to explore outcomes in patients with acute kidney injury (AKI) and sepsis submitted to continuous renal replacement therapy (CRRT) with Oxiris™.

Objectives:

Describe the experience and outcomes in patients with sepsis and AKI treated receiving CRRT with the adsorption membrane filter Oxiris™

DETAILED DESCRIPTION:
Study Background & Rationale:

Acute kidney injury (AKI) is common in patients with sepsis, occurring in 5-50%. It happens in the context of a critical illness requiring intensive care. Fifteen percent require renal replacement therapy as supportive therapy until the kidneys recover. Membrane-coated filters, such as Oxiris™, promote high filtration clearance of uremic toxins, but additionally removal of inflammatory mediators and bacterial liposaccharide (LPS) . Even though this potential mechanism should be expected to benefit septic and AKI patients, results have not been uniform.

The investigators´ group has been prescribing CRRT for AKI treatment for the last 20 years, having performed more than 20 thousand procedures. The investigators´ group experience with Oxiris™ filter in CRRT started in 2018. The objective of the study is to describe the clinical operational management of CRRT with this kind of filter and to explore patients' outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Adults (>18 years)
* Diagnosis of AKI (KDIGO stage 3)
* Diagnosis of sepsis of any cause

Exclusion Criteria:

* COVID19 diagnosis

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with sepsis and acute kidney injury treated receiving continuous renal replacement therapy with the adsorption membrane filter Oxiris
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2023-12-08 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Mortality observed and estimated by predictive indexes | Through study completion, an average of 5 years
  In-hospital mortality observed and estimated by the predictive index (SAPS III) during the hospitalization which developed AKI and need CRRT with Oxiris

SECONDARY OUTCOMES:
Management of hemodynamic drugs during CRRT | Through study completion, an average of 5 years
  Daily dosage of hemodynamic active drugs (mg/day) during the hospitalization which developed AKI and need CRRT with Oxiris
Hemorrhagic complications during CRRT | Through study completion, an average of 5 years
  Occurrence of hemorrhagic events during the hospitalization which developed AKI and need CRRT with Oxiris
CRRT circuit life-time | Through study completion, an average of 5 years
  Days of CRRT circuit with Oxiris utilization, during the hospitalization which developed AKI and need CRRT with Oxiris
CRRT dependence | Through study completion, an average of 5 years
  Time in days on CRRT need, during the hospitalization which developed AKI and need CRRT with Oxiris
Initial renal function recovery | Through study completion, an average of 5 years
  Time in days to urinary debt >1L/day, during the hospitalization which developed AKI and need CRRT with Oxiris
Length of hospital stay | Through study completion, an average of 5 years
  Length of hospital stay in days of hospitalization which developed AKI and need CRRT with Oxiris
Renal function recovery in medium term | At 30 days after hospital admission in which participants developed AKI
  Renal function by creatinine levels (mg/dl) at 30 days after hospital admission of the hospitalization which developed AKI and need CRRT with Oxiris
Renal function recovery at discharge | Through study completion, an average of 5 years
  Renal function by creatinine levels (mg/dl) at discharge of the hospitalization which developed AKI and need CRRT with Oxiris
Dialysis dependence in long term | Through study completion, an average of 5 years
  Dialysis dependence at discharge of the hospitalization which developed AKI and need CRRT with Oxiris

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth R Maccariello, MD, PhD, Principal Investigator — Nefro Consultoria de Doenças Renais
Locations (1):
- Nefro Consultoria de Doenças Renais, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Hoste EAJ, Kellum JA, Selby NM, Zarbock A, Palevsky PM, Bagshaw SM, Goldstein SL, Cerda J, Chawla LS. Global epidemiology and outcomes of acute kidney injury. Nat Rev Nephrol. 2018 Oct;14(10):607-625. doi: 10.1038/s41581-018-0052-0. PMID 30135570
- [Result] Malard B, Lambert C, Kellum JA. In vitro comparison of the adsorption of inflammatory mediators by blood purification devices. Intensive Care Med Exp. 2018 May 4;6(1):12. doi: 10.1186/s40635-018-0177-2. PMID 29728790
- [Result] Peerapornratana S, Manrique-Caballero CL, Gomez H, Kellum JA. Acute kidney injury from sepsis: current concepts, epidemiology, pathophysiology, prevention and treatment. Kidney Int. 2019 Nov;96(5):1083-1099. doi: 10.1016/j.kint.2019.05.026. Epub 2019 Jun 7. PMID 31443997
- [Result] Maccariello E, Soares M, Valente C, Nogueira L, Valenca RV, Machado JE, Rocha E. RIFLE classification in patients with acute kidney injury in need of renal replacement therapy. Intensive Care Med. 2007 Apr;33(4):597-605. doi: 10.1007/s00134-007-0535-0. Epub 2007 Feb 20. PMID 17310365
- [Result] Maccariello E, Valente C, Nogueira L, Bonomo H, Ismael M, Machado JE, Baldotto F, Godinho M, Valenca R, Rocha E, Soares M. SAPS 3 scores at the start of renal replacement therapy predict mortality in critically ill patients with acute kidney injury. Kidney Int. 2010 Jan;77(1):51-6. doi: 10.1038/ki.2009.385. PMID 19812539
- [Result] Bouchard J, Acharya A, Cerda J, Maccariello ER, Madarasu RC, Tolwani AJ, Liang X, Fu P, Liu ZH, Mehta RL. A Prospective International Multicenter Study of AKI in the Intensive Care Unit. Clin J Am Soc Nephrol. 2015 Aug 7;10(8):1324-31. doi: 10.2215/CJN.04360514. Epub 2015 Jul 20. PMID 26195505